CLINICAL TRIAL: NCT06316726
Title: The Effectiveness of Two Nursing Programs on the Surgery-Related Pressure Injury in Surgery Patients
Brief Title: The Effectiveness of Two Nursing Programs on the Surgery-related Pressure Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202100409A3
Record Dates: First submitted 2024-02-29; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2021-05

CONDITIONS: Pressure Injury; Surgery
Keywords: surgery-related pressure injury; incidence; grade; sites; time
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: The experimental group was randomly assigned by block to receive intervention A (full bed silicone mattress plus other measures), and the control group received intervention B (full bed silicone mattress plus usual care).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention A (Active Comparator): full bed silicone mattress plus other measures
  Interventions: Combination Product: full bed silicone mattress plus other measures
- intervention B (No Intervention): full bed silicone mattress plus usual care

INTERVENTIONS:
Combination Product: full bed silicone mattress plus other measures — full bed silicone mattress plus put silicone pads on the head and shoulders, cotton rolls wraps bony prominence (elbows and heels), petrissage every two hours on shoulders to fingers and lower legs to heels, change location of ankle pads, use round gel full of air sit pad, a pillow on the knees
  Arms: intervention A

SUMMARY:
Introduction: This study was to compare the differences in the incidence, grade, and time of surgery-related pressure injuries between the two interventions; and describe the locations of surgery-related pressure injuries between the two interventions.

Methods: This study adopted a true experimental research design with a convenience sampling method from the operating rooms of a teaching hospital in a northern region. The experimental group was randomly assigned by block to receive intervention A (full bed silicone mattress plus other measures), and the control group received intervention B (full bed silicone mattress plus usual care). Measurements include basic personal attributes, risk factors, grade, time, and location of occurrence related to surgery-related pressure injuries.

ELIGIBILITY:
Inclusion Criteria:

* 20 and more years old
* Over 4 hours lying flat on the operating table (eg., orthognathic surgery, microtia reconstruction surgery, etc.)
* Those who are conscious clearly and can communicate in Mandarin and Taiwanese
* Those with agree to participate in this study

Exclusion Criteria:

* Those whose skin is red, swollen, hot, painful, redness, rash, purple spots, bruising, scaly skin, damaged, etc.
* Refuse to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
the occurrence of surgery-related pressure injuries | baseline, pre-surgery; every two hours during the surgery till ten hours; and post-surgery to the 2nd day after surgeryl
  incidence, grade, site, and time of surgery-related pressure injuries

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chu Tsai, MN, Study Director — Nursing Department of Taoyuan Chang Gung Memorial Hospital
Locations (1):
- Taoyuan Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nixon J, McElvenny D, Mason S, Brown J, Bond S. A sequential randomised controlled trial comparing a dry visco-elastic polymer pad and standard operating table mattress in the prevention of post-operative pressure sores. Int J Nurs Stud. 1998 Aug;35(4):193-203. doi: 10.1016/s0020-7489(98)00023-6. PMID 9801935
- [Result] Feuchtinger J, de Bie R, Dassen T, Halfens R. A 4-cm thermoactive viscoelastic foam pad on the operating room table to prevent pressure ulcer during cardiac surgery. J Clin Nurs. 2006 Feb;15(2):162-7. doi: 10.1111/j.1365-2702.2006.01293.x. PMID 16422733
- [Result] Sewchuk D, Padula C, Osborne E. Prevention and early detection of pressure ulcers in patients undergoing cardiac surgery. AORN J. 2006 Jul;84(1):75-96. doi: 10.1016/s0001-2092(06)60100-2. PMID 16881492
- [Result] Donnelly J, Winder J, Kernohan WG, Stevenson M. An RCT to determine the effect of a heel elevation device in pressure ulcer prevention post-hip fracture. J Wound Care. 2011 Jul;20(7):309-12, 314-8. doi: 10.12968/jowc.2011.20.7.309. PMID 21841719
- [Result] Oliveira KF, Pires PDS, De-Mattia AL, Barichello E, Galvao CM, Araujo CA, Barbosa MH. Influence of support surfaces on the distribution of body interface pressure in surgical positioning. Rev Lat Am Enfermagem. 2018 Nov 29;26:e3083. doi: 10.1590/1518-8345.2692.3083. PMID 30517574
- [Result] Joseph J, McLaughlin D, Darian V, Hayes L, Siddiqui A. Alternating Pressure Overlay for Prevention of Intraoperative Pressure Injury. J Wound Ostomy Continence Nurs. 2019 Jan/Feb;46(1):13-17. doi: 10.1097/WON.0000000000000497. PMID 30601427
- [Result] Neo TG, Koo SH, Chew STH, Png GK, Lacuesta MJ, Wu MYL, Tay RYC, Singh PA, Chandran R. A randomized controlled trial to compare the interface pressures of alternating pressure overlay with gel pad versus gel pad alone during prolonged surgery. J Tissue Viability. 2021 May;30(2):222-230. doi: 10.1016/j.jtv.2021.02.003. Epub 2021 Feb 6. PMID 33612359
- [Result] Ahmad B, Rubio-Sefati M, Yacob MM. Incidence and risk factors for pressure injuries in patients who have undergone vascular operations: a scoping review. Eur J Med Res. 2023 Feb 13;28(1):77. doi: 10.1186/s40001-023-01036-3. PMID 36782315
- [Result] Chen HL, Chen XY, Wu J. The incidence of pressure ulcers in surgical patients of the last 5 years: a systematic review. Wounds. 2012 Sep;24(9):234-41. PMID 25874704